CLINICAL TRIAL: NCT03410576
Title: Comparison of the Perioperative Time Course of Matrix Metalloproteinase-9 (MMP-9) and Its Inhibitor (TIMP-1) During Carotid Artery Stenting (CAS) and Carotid Endarterectomy (CEA)
Brief Title: Perioperative Time Course of MMP-9 and Its Inhibitor During Carotid Artery Stenting and Carotid Endarterectomy
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Gábor László Woth, Principal investigator, University of Pecs
Other Study IDs: 5016
Record Dates: First submitted 2018-01-06; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Carotid Stenosis; Ischemia Reperfusion Injury
Keywords: Matrix metalloproteinase; Carotid artery stenting; Carotid endarterectomy
MeSH Terms: conditions — Carotid Stenosis; Reperfusion Injury | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carotid artery stenting: Patients undergo carotid artery stenting.
  Interventions: Procedure: Carotid artery stenting
- Carotid endarterectomy: Patients receive elective carotid endarterectomy.
  Interventions: Procedure: Carotid endarterectomy

INTERVENTIONS:
Procedure: Carotid artery stenting — Patient undergo elective carotid artery stenting. In this patient group blood sampling was performed at three time points: T1, at the time of the insertion of the arterial line; T2, 60 min after stent insertion; and T3: the first postoperative morning.
  Groups: Carotid artery stenting
Procedure: Carotid endarterectomy — Patient undergo elective carotid endarterectomy. Group samples were collected at the following four time points: T1, at the time of the insertion of the arterial line; T2, 60 min after cross-clamp release; T3, the first postoperative morning; and T4, the third postoperative morning. A matched subgroup of patients from the previously obtained data served as a historical control.
  Groups: Carotid endarterectomy

SUMMARY:
The aim was the comparison of the perioperative time courses of matrix metalloproteinase-9 (MMP-9) and its inhibitor (TIMP-1) during elective carotid artery stenting (CAS). The investigators used a matched, historical carotid endarteriectomy group as controls. Blood samples at four time points: T1: preoperative; T2: 60 minutes after stent insertion; T3: first postoperative morning; and T4: third postoperative morning. Plasma was isolated from heparin anticoagulated blood samples by low speed centrifugation at 4 °C, and stored at -80 °C until analyzed in a single batch at the end of the study. Plasma concentrations of MMP-9 and TIMP-1 were expressed as ng/ml.

ELIGIBILITY:
Inclusion Criteria:

elective carotid artery surgery

Exclusion Criteria:

Malignant diseases, inflammatory and systemic autoimmune disorders, psychiatric disorders and previous debilitating stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed carotid artery stenosis
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Plasma MMP-9 concentrations | 4 days
  Plasma is isolated from heparin-anticoagulated blood samples by low speed centrifugation at 4 °C. MMP-9 levels were measured with quantitative sandwich enzyme-linked immunosorbent assay.
Plasma TIMP-1 concentrations | 4 days
  Plasma is isolated from heparin-anticoagulated blood samples by low speed centrifugation at 4 °C. TIMP-1 levels were measured with quantitative sandwich enzyme-linked immunosorbent assay.

SECONDARY OUTCOMES:
MMP-9/TIMP-1 ratio | 4 days
  MMP-9/TIMP-1 is calculated from the measured plasma MMP-9 and TIMP-1 concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Gábor Woth, MD, PhD, Principal Investigator — Department of Anaesthesiology and Intensive Therapy, Medical School, University of Pécs; Bálint Nagy, MD, PhD, Principal Investigator — Department of Anaesthesiology and Intensive Therapy, Medical School, University of Pécs; Diana Mühl, MD, PhD, Study Director — Department of Anaesthesiology and Intensive Therapy, Medical School, University of Pécs; János Lantos, PhD, Principal Investigator — Department of Surgical Research and Techniques, Medical School, University of Pécs,; Ferenc Kövér, MD, Principal Investigator — Department of Neurosurgery, Medical School, University of Pécs,; Lajos Bogár, MD, DsC, Principal Investigator — Department of Anaesthesiology and Intensive Therapy, Medical School, University of Pécs
Locations (1):
- Department of Anaesthesiology and Intensive Therapy, Medical School, University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagy B, Woth G, Merei A, Nagy L, Lantos J, Menyhei G, Bogar L, Muhl D. Perioperative time course of matrix metalloproteinase-9 (MMP-9), its tissue inhibitor TIMP-1 & S100B protein in carotid surgery. Indian J Med Res. 2016 Feb;143(2):220-6. doi: 10.4103/0971-5916.180212. PMID 27121520
- [Derived] Merei A, Nagy B, Woth G, Lantos J, Kover F, Bogar L, Muhl D. Comparison of the perioperative time courses of matrix metalloproteinase-9 (MMP-9) and its inhibitor (TIMP-1) during carotid artery stenting (CAS) and carotid endarterectomy (CEA). BMC Neurol. 2018 Aug 29;18(1):128. doi: 10.1186/s12883-018-1133-1. PMID 30157791